CLINICAL TRIAL: NCT07094529
Title: The Feasibility of Personalized Hypoglycemia Outpatient Treatment for People Living With Type 2 Diabetes Mellitus
Brief Title: Personalized Hypoglycemia Outpatient Treatment - a Feasibility Study
Acronym: PHOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250297-01H
Record Dates: First submitted 2025-07-21; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes (T2DM); Hypoglycemia (Diabetic)
Keywords: hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recumbent Exercise Bike to induce mild hypoglycemia (Experimental): The participant rides the recumbent exercise bike at their preferred speed and records the distance travelled until there is onset of mild hypoglycemia.
  Interventions: Behavioral: Recumbent Exercise Bike to induce mild hypoglycemia
- Delaying food to induce mild hypoglycemia (Experimental): At the study visit, in front of the study nurse, the participant takes their usual clinical care dose of sulfonylurea or basal insulin. If the participant's usual clinical care includes insulin with a rapid-acting component, then its dose is reduced based on the study protocol.
  Interventions: Behavioral: Delaying food to induce mild hypoglycemia,

INTERVENTIONS:
Behavioral: Recumbent Exercise Bike to induce mild hypoglycemia — The participant rides the recumbent exercise bike at their preferred speed and records the distance travelled until there is onset of mild hypoglycemia, determined by capillary blood glucose test result 3.0 to 3.8 mmmol/L.
  Based on each participant's own experience with hypoglycemia treatment or their preferences, the participant can choose one of 4 simple carbohydrate treatment quantities: 8 grams, 16 grams, 20 grams, 32 grams
  The participant can choose one of 4 capillary blood glucose recheck times: 15 minutes, 20 minutes, 25 minutes, 30 minutes.
  Arms: Recumbent Exercise Bike to induce mild hypoglycemia
Behavioral: Delaying food to induce mild hypoglycemia, — At the study visit, in front of the study nurse, the participant takes their usual clinical care dose of sulfonylurea or basal insulin. If the participant's usual clinical care includes insulin with a rapid-acting component, then its dose is reduced based on the study protocol.
  No food intake (water is allowed) until there is onset of mild hypoglycemia, determined by a capillary blood glucose test result 3.0 to 3.8 mmol/L.
  Based on each participant's own experience with hypoglycemia treatment or their preferences, the participant can choose one of 4 simple carbohydrate treatment quantities: 8 grams, 16 grams, 20 grams, 32 grams
  The participant can choose one of 4 capillary blood glucose recheck times: 15 minutes, 20 minutes, 25 minutes, 30 minutes.
  Arms: Delaying food to induce mild hypoglycemia

SUMMARY:
This study will offer two study interventions designed to bring on a mild low blood sugar (capillary blood glucose result 3.0 to 3.8 mmol/L), in order to study the effectiveness of each study participant's personal choice of treatment and first recheck time.

The two study interventions that the participant can choose to complete (one or both interventions).

Based on each participant's own experience with hypoglycemia treatment or their preferences, the participant can choose one of 4 simple carbohydrate treatment quantities, and choose one of 4 capillary blood glucose recheck times.

DETAILED DESCRIPTION:
The two study interventions that the participant can choose to complete (one or both interventions):

Study intervention A: Ride a recumbent exercise bike at participant's own desired speed, until onset of capillary blood glucose showing mild low blood glucose (hypoglycemia).

Study intervention B: Delay food intake after the participant brings and takes their routine clinical care prescribed medication(s) that decrease the blood glucose level. The participant brings in their medication(s) including sulfonylurea or insulin(s) as applicable to the study visit. In front of the study nurse, the participant takes these medication(s) at the same dose or reduced dose as defined in the study protocol. The participant is monitored until capillary blood glucose reaches the mild low blood glucose (hypoglycemia) level of 3.0 to 3.8 mmol/L.

Based on each participant's own experience with hypoglycemia treatment or their preferences, the participant can choose one of 4 simple carbohydrate treatment quantities: 8 grams, 16 grams, 20 grams, 32 grams

The participant can choose one of 4 capillary blood glucose recheck times: 15 minutes, 20 minutes, 25 minutes, 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, an individual must meet all of the following criteria:

  1. Consent provided
  2. Age >= 18 years.
  3. Diagnosed as type 2 diabetes mellitus.
  4. Type 2 diabetes medications include at least one of the following for at least one month prior to entering the study: sulfonylurea or insulin of any type.

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:

  1. Diagnosed as another form of diabetes mellitus.
  2. Has a history of hypoglycemia unawareness.
  3. Had a hypoglycemia event, defined as capillary blood glucose < 3.9 mmol/L within 24 hours prior to the study visit booking time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
To determine feasibility to recruit an average of 8 patients per month at the study site (The Ottawa Hospital Diabetes clinics) for study protocol performance. | 12 months
  Average number of patients recruited per month is determined by 60 patients (the target recruitment number) for each study intervention, divided by the number of months that it took to complete the recruitment.

SECONDARY OUTCOMES:
To assess the percentage hypoglycemia resolution for people living with type 2 diabetes based on their personalized choice of treatment and first recheck time. | 12 months
  Percentage hypoglycemia resolution with respect to grams of simple carbohydrates that participant chose, and first recheck time that participant preferred.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Sun, MD MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No